CLINICAL TRIAL: NCT02349646
Title: A Post Market Cohort With the Commercially Available Spinal Modulation Neurostimulator System for the Management of Peripheral Neuropathy
Brief Title: A Post Market Cohort With the Spinal Modulation Neurostimulator System in Peripheral Neuropathy
Status: Terminated | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-SMI-2012
Record Dates: First submitted 2015-01-07; First posted 2015-01-29 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated subjects: All subjects recruited and treated with the Axium neurostimulator
  Interventions: Device: Implantation with the commercially available Axium neurostimulator

INTERVENTIONS:
Device: Implantation with the commercially available Axium neurostimulator

SUMMARY:
10-SMI-2012 is a post market observational, questionnaire based study to assess the effectiveness of the commercially available Axium neurostimulator in the management of peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Peripheral neuropathy for at least 6 months
4. Failed conservative treatments for chronic pain including but not limited to pharmacological therapy, physical therapy and interventional pain procedures for chronic pain
5. Average baseline pain rating of 60 mm on the Visual Analog Scale in the primary region of pain
6. In the opinion of the Investigator, the subject is psychologically appropriate for the implantation for an active implantable medical device
7. Subject is able to provide written informed consent

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
4. Subject has had radiofrequency treatment of an intended target dorsal root ganglion within the past 3 months
5. Subject currently has an active implantable device including implanted cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Subjects currently has an active infection
8. Subject has, in the opinion of the Investigator, a medical comorbidity that contraindicates placement of an active medical device
9. Subject has participated in another clinical investigation within 30 days that may confound the outcomes of the current study as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peripheral Neuropathy Patients
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich Heine Universität Düsseldorf, Düsseldorf, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Axium DRG Neurostimulator: All subects implanted with intent to treat with the Axium DRG Neurostimulator
Period: Overall Study
Arm/Group | Axium DRG Neurostimulator
Started | 33
Received Trial System | 24
Receive Permanent System | 27
Completed | 16
Not Completed | 17

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with the Axium Neurostimulator
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 51 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity for Overall Pain From Pre-treatment Baseline
Description: The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum pain) to 10 (maximum pain).
Time Frame: Baseline, 3, 6 and 12-Month Visits
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subjected Treated With the Permanent Implantable Axium System: All subjects treated with the Axium implantable neurostimulator
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 33
units on a scale
  Baseline | 7.4 (1.7)
  3-Month Visit: number analyzed (Participants) | 23
  3-Month Visit | 4.0 (2.6)
  6-Month Visit: number analyzed (Participants) | 20
  6-Month Visit | 3.4 (2.5)
  12-Month Visit: number analyzed (Participants) | 16
  12-Month Visit | 3.8 (2.5)

2. Primary Outcome: Percentage of Subjects With at Least 50% Pain Reduction
Description: Percent of subjects with at least a 50% reduction. The Visual Analog Scale (VAS) is self-administered instrument assessing average pain intensity. Subjects rated their pain on a horizontal line, 10 cm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher pain level. The values range from 0 (minimum) to 10 (maximum).
Time Frame: 3, 6 and 12-Month Visits
Population: Differences in participants over time is due to early withdrawals and missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Subjected Treated With the Permanent Implantable Axium System
Number analyzed (Participants) | 23
Participants
  3-Month Visit | 13
  6-Month Visit: number analyzed (Participants) | 20
  6-Month Visit | 14
  12-Month Visit: number analyzed (Participants) | 16
  12-Month Visit | 8

ADVERSE EVENTS:
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 8/33
Other Adverse Events (participants affected / at risk) | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=33)
IPG Pocket Pain due to IPG displacement to ventral (Product Issues) | 1 (1)
Loss of Stimulation (Product Issues) | 1 (1)
Conus cauda syndrome (Nervous system disorders) | 1 (1)
CSF leak (Injury, poisoning and procedural complications) | 1 (1)
Infection at IPG site (Infections and infestations) | 1 (1)
Leriche's syndrome (Vascular disorders) | 1 (1)
Loss of bladder control, sensational numbness, coordination problem right arm (Injury, poisoning and procedural complications) | 1 (1)
Nausea and headache (Injury, poisoning and procedural complications) | 1 (1) — This Adverse Events was monitored/assessed in such a manner that the specific Adverse Event Terms cannot be separated.
Suicide Attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=33)
Loss of Stimulation (Product Issues) | 3 (3)
Hematoma (Vascular disorders) | 1 (1)
Overstimulation (Product Issues) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days